CLINICAL TRIAL: NCT03157791
Title: Addition of Oral Simethicone to Bowel Preparation in Colonoscopy
Brief Title: Simethicone and Bowel Preparation in Colonoscopy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: University of Manitoba (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Diagnostic
Other Study IDs: B2017:056
Record Dates: First submitted 2017-05-15; First posted 2017-05-17 (Actual); Last update posted 2018-05-23 (Actual); Status verified 2017-05

CONDITIONS: Colonoscopy; Bowel Preparation
Keywords: simethicone
MeSH Terms: interventions — Simethicone; Capsules

STUDY DESIGN:
Who Masked: Investigator, Outcomes Assessor
Masking Description: The endoscopist and endoscopy nurse will not know to which treatment arm the patient belongs as only the interviewing nurse will have taken down this information. This information does not travel with the patient to the endoscopy room. The patient is also instructed to not reveal to the endoscopist or endoscopy nurse if he or she has taken simethicone or not.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Simethicone with Bowel Prep (Experimental): Group A will receive 2 simethicone tablets (180mg each) so that one tablet is taken at the same time as each bowel preparation dose.
  Interventions: Drug: Simethicone 180Mg Cap
- Control (No Intervention): Group B will receive no simethicone tablets.

INTERVENTIONS:
Drug: Simethicone 180Mg Cap — Simethicone Group A will take a total of 360mg prior to colonoscopy of Simethicone 180Mg Cap.
  Other Names: Gas-X
  Arms: Simethicone with Bowel Prep

SUMMARY:
This Clinical Trial is being conducted to study the effect of oral simethicone on the presence of bubbles during colonoscopy. The purpose of this study is to find out what effects (good and bad) the addition of oral simethicone to bowel preparation has on the ability to visualize the colon mucosa (bowel) during colonoscopy.

DETAILED DESCRIPTION:
Evaluation of the lower gastrointestinal (GI) tract by colonoscopy is now considered the gold standard and its use is on the rise in all GI units. Clean bowel preparation is a mandatory part of the procedure in order to visualize the bowel mucosa to determine pathology and provide therapeutic intervention safely if needed.

Colon lavage preparations have been effective in improving visibility of the colon and are well tolerated. Split dose bowel preparation regimens have been developed and adapted in order to optimize patient comfort and provide adequate cleanliness .

These bowel preparations address issues regarding the feculent residual material, however bubbles lining the mucosa remain a problem in attempting to visualize the colon mucosa. About 30% of adequately prepared bowels are now affected with mucosa lined with bubbles . The bubbles limit evaluation of the entire bowel, requiring more time to clean the bowel and possibly missing pathology such as small, flat sessile, serrated polyps, small apthous ulcers for crohns and many other pathologies.

Simethicone is a mixture of polydimethylsiloxane and hydrated silica gel and works by reducing surface tension of air bubbles, allowing small bubbles to coalesce to form larger bubbles allowing the air to pass as belching or flatulence. This makes simethicone an ideal antifoaming agent that has been used in all age groups to reduce bloating, abdominal discomfort, and abdominal pain.

In the past, use of simethicone in the irritant fluid has been used to wash away the bubbles, however there has been recent concern with scope manufacturers advising that simethicone not to be used routinely because of simethicone settling in the irrigation channel. This causes a concerning biofilm in the endoscope.

Use of oral simethicone instead of liquid simethicone through the endoscope as an adjuvant to the bowel preparation to reduce bubbles/foam has not been adopted widely due to lack of knowledge and literature available and the project's ability to secure funding. This project aims to compare the amount of bubbles and colon mucosa visibility between patients who ingested oral simethicone with bowel preparation and those who did not to evaluate the use of oral simethicone in future colonoscopies.

All patients who are referred to undergo colonoscopy are booked centrally in the GI Unit at the Brandon Regional Health Centre (BRHC) and are given instructions regarding bowel preparation and procedure time by the booking department. All patients including those not involved in research are instructed and scheduled in the same manner.

About a month prior to procedure all patients are sent bowel preparation instructions, procedure time and colonoscopy information. A letter explaining the study and requesting participation will be included with this information.

All patients are instructed to call the GI Unit 5 days prior to their procedure to confirm. At this time patients will be asked to participate in the study by the Clinical Resource Nurse (CRN) or CRN delegate.

Treatment group is determined by the number on each consent form. This number will be referenced with the master list to determine if the patient is in Group A or Group B. Participants will all be advised to not speak to the endoscopist about whether they have taken simethicone tablets or not. If participants were allotted to group A but present on the day of the procedure without having taking simethicone they will be excluded from the study.

On the day patients present to the GI unit for their colonoscopy they will undergo the same process as a participant not in the study. Participants will present to the interview desk. The patient will be reminded to not tell any physician or nurse other than the interview nurse. The interviewing nurse will ask the patient if they ingested the simethicone and if so what dosage and what brand of tablets. This will be noted on the simethicone ingestion form that will be placed in an envelope and in the appropriate folder in accordance with the treatment group to which the participant belongs. The interviewing nurse will then proceed with the regular intake form.

The endoscopy room will have the Boston Bowel Preparation Scale and the Bubble Scale labeled with appropriate participant number. The endoscopist will complete these forms once the procedure is finished and will be blinded as to which group the patient belongs. Once completed by the endoscopy nurse a photocopy of the Endoscopy Room Quality Indicators form will be placed with the participant folder with the identifying information blacked out and replaced with the participant number. All the completed forms will be collated and placed in a sealed envelope by the recovery room nurse and placed in the appropriate folder in accordance with the treatment group to which the participant belongs.

The amount of bubbles will be compared between Group A (simethicone) and Group B (no simethicone) using a chi square analysis with a statistical significance value of p=0.5. The same will be done for bowel cleanliness using the Ottawa stool scale.

ELIGIBILITY:
Inclusion Criteria:

* Patients receiving colonoscopy who are within 30km of Brandon Manitoba and no other exclusion criteria

Exclusion Criteria:

* inability to provide informed consent, under 18 years old, inpatient, pregnancy, known hypersensitivity to simethicone, or excessive language barriers.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 471 (Actual)
Dates: Start 2017-07-05 (Actual); Primary Completion 2017-11-26 (Actual); Study Completion 2017-11-26 (Actual)

PRIMARY OUTCOMES:
Bubble Scale Score | Will be completed immediately after colonoscopy is completed
  The scale grades the amount of bubbles present in the colon from 0 (none) to 3 (severe)

SECONDARY OUTCOMES:
Ottawa Stool Scale | Will be completed immediately after colonoscopy is completed
  The scale grades the degree of bowel preparation from 0 (no preparation) to 3 (entire colon mucosa seen well)

CONTACTS AND LOCATIONS:
Overall Officials: Melissa Towle, RN, Study Director — Brandon Regional Health Centre; Charlenn Skead, BA, Study Director — University of Manitoba
Locations (1):
- Brandon Regional Health Centre, Brandon, Manitoba, Canada

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Goldman J, Reichelderfer M. Evaluation of rapid colonoscopy preparation using a new gut lavage solution. Gastrointest Endosc. 1982 Feb;28(1):9-11. doi: 10.1016/s0016-5107(82)72956-6. PMID 7056467
- [Background] Martel M, Barkun AN, Menard C, Restellini S, Kherad O, Vanasse A. Split-Dose Preparations Are Superior to Day-Before Bowel Cleansing Regimens: A Meta-analysis. Gastroenterology. 2015 Jul;149(1):79-88. doi: 10.1053/j.gastro.2015.04.004. Epub 2015 Apr 8. PMID 25863216
- [Background] Matro R, Tupchong K, Daskalakis C, Gordon V, Katz L, Kastenberg D. The effect on colon visualization during colonoscopy of the addition of simethicone to polyethylene glycol-electrolyte solution: a randomized single-blind study. Clin Transl Gastroenterol. 2012 Nov 29;3(11):e26. doi: 10.1038/ctg.2012.16. PMID 23238113
- [Background] Parikh VA, Khanduja KS. Use of simethicone during colonoscopy. Dis Colon Rectum. 1995 Sep;38(9):1007-8. doi: 10.1007/BF02049743. No abstract available. PMID 7656734
- [Background] Ofstead CL, Wetzler HP, Johnson EA, Heymann OL, Maust TJ, Shaw MJ. Simethicone residue remains inside gastrointestinal endoscopes despite reprocessing. Am J Infect Control. 2016 Nov 1;44(11):1237-1240. doi: 10.1016/j.ajic.2016.05.016. Epub 2016 Aug 3. PMID 27497824